CLINICAL TRIAL: NCT02783989
Title: A Single-center, Crossover, Randomized and Controlled Nutritional Intervention Clinical Trial. A Nutritional Intervention Study
Brief Title: Effects on Cardiovascular Risk Factors of the Endogenous Hydroxytyrosol Generation After the Combined Intake of Wine and Tyrosol in Humans
Acronym: DOPET3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, Pharm D, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IMIMFTCLFT/DOPET/3
Record Dates: First submitted 2016-05-11; First posted 2016-05-26 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Disease
Keywords: Endothelial function; Inflammation; Genes related to vascular risk
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — 4-hydroxyphenylethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- White wine (Active Comparator): Two glasses of a market white wine (2x135 mL, 13º), each (135 mL) equivalent to 14 g of ethanol (in case of women only one glass, 135 mL), being the daily dose of 28 g (14 g in women). It is estimated that wine will contain about 8-9 mg/l of tyrosol. Therefore the dose of tyrosol ingested in two glasses would be 2-2.5 mg (1-1.25 mg in women).
  Interventions: Other: white wine
- White wine plus tyrosol capsules (Experimental): Two glasses of white wine (2x135 mL, 13º), each (135 mL) equivalent to 14 g of ethanol (in case of women only one glass, 135 mL), being the daily dose of 28 g (14g in women), in combination with capsules of 25 mg of TYR (each one to be ingested with a glass of wine), two capsules along the day for men (at lunch and at dinner) and one for woman (at lunch).
  Interventions: Other: white wine; Dietary Supplement: tyrosol
- Water (No Intervention): Drinking water along with meals

INTERVENTIONS:
Other: white wine — A dietary beverage: a market white wine, 13º alcohol
  Arms: White wine; White wine plus tyrosol capsules
Dietary Supplement: tyrosol — tyrosol in capsules
  Arms: White wine plus tyrosol capsules

SUMMARY:
The present study will assess whether the beneficial effects of a market moderate-alcohol drinking in the form of white wine in humans could be derived from the endogenous formation of hydroxytyrosol (also known DOPET), a potent dietary anti-inflammatory and antioxidant molecule.

DETAILED DESCRIPTION:
Epidemiological studies support that light to moderate alcohol drinking (10-20g per day), may reduce the risk of cardiovascular disease (CVD), stroke, dementia, depression, and all-cause mortality. In addition, moderate red wine consumption has recently shown to be inversely associated with a decline in global cognitive function and the domains of memory and flexibility. The claimed beneficial effects of the Mediterranean diet include prevention of several age-related dysfunctions including cardiovascular and neurodegenerative diseases. These effects have been related to the protection against cognitive decline associated with aging and disease by a number of polyphenols found in red wine and virgin olive oil. Neurodegenerative diseases, as all chronic degenerative diseases, are linked to inflammation and its inter-twined phenomena: the oxidation and the oxidative damage. The interrelationship among chronic degenerative diseases is also evidenced by the fact that vascular (cardiovascular) risk factors are associated to cognitive decline, and these vascular factors are currently the only known modifiable risk factors for Alzheimer disease.

There is evidence suggesting that DOPET, also known as hydroxytyrosol (HOTYR), has a role in the cardioprotective and neuroprotective properties of wine. It is a phenolic compound present in virgin olive oil and wine, and it is a potent dietary anti-inflammatory and antioxidant molecule. Biological effects of HOTYR may explain in part some of the beneficial effects for human health that have been credited to moderate ethanol intake (in form of wine).

The present project is not intended to provide support for the clinical use of moderate- dose alcohol as a treatment modality for CVD risk patients. Nevertheless, it will investigate a novel mechanism of action that may explain in part beneficial health effects associated to moderate alcohol consumption. This novel mechanism of action is mediated by compounds that at mid/long-term run are susceptible of a pharmaceutical and/or nutraceutical food development.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and accepting the study procedures and signing the informed consent.
2. Male and female volunteers aged 50 to 80 years.
3. Participants with at least three major cardiovascular risk factors, including:

   * current smoking (>1 cig/day during the last month)
   * hypertension ≥140/90 mmHg or antihypertensive medication
   * low-density lipoprotein (LDL)-cholesterol >130 mg/dl or lipid-lowering therapy
   * low high-density lipoprotein (HDL)-cholesterol ≤40 mg/dl in men or ≤50 mg/dl in women
   * overweight/obesity (body mass index≥25 kg/m2)
   * a family history of premature coronary heart disease (CHD).
4. Clinical diagnosis of type 2 diabetes.
5. Clinical history and physical examination demonstrating no organic or psychiatric disorders.
6. The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
7. Subjects socially drinking and who had ingested wine at least once.
8. Acceptance of following a controlled diet with a moderate content of antioxidants along the study, in which time it will be not permitted the consumption of wine/champagne (except in the framework of treatment conditions in the clinical trial) or other alcoholic drinks (beer, spirits…), but it will be allowed a maximum of:

   (i) Vegetables (including pulses): one serving (small dish)/day; (ii) Fruits (or juices): 2 pieces/day; (iii) Commercial olive oil: maximum 25 mL/day; (iv) Drinks containing xanthines (coffee, tea, cola, energy drinks…): maximum 3 cups/day; (v) Chocolate: maximum one piece (small, 15 gr)/day; (vi) Nuts: maximum 30 g (a small handful)/week; and (vii) Fish: maximum 3 times per week (150g/serving).

Exclusion Criteria:

1. Not meeting the inclusion criteria.
2. Participants with BMI >40kg/m2
3. Participants who intake antioxidant supplements.
4. Participants with multiple allergies or intestinal diseases.
5. Participants who follow special diets (vegetarian and vegan diets included).
6. Participants with any condition limiting their mobility, making study visits impossible or worsening the adherence to the treatments.
7. Participants with history of hypersensitivity or intolerance to ethanol.
8. Ethanol users of >80 g/d (v) and illicit drug users.
9. Illiteracy.
10. Participants with an acute infection or inflammatory process in the last three months (may be included if the episode developed prior to 3 months).
11. Participants with history of previous cardiovascular disease (coronary heart disease or stroke)
12. Participants taking medication with sedative effects or interacting with ethanol.
13. Participation in other clinical trials with drugs in the previous 12 weeks

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Metabolic: changes in hydroxytyrosol generation | change from baseline at 4 weeks
  Hydroxytyrosol generation from tyrosol ingestion in urine (24 hours urine collection)
Vascular effects: changes in endothelial function | change from baseline at 4 weeks
  It will be measured in the morning by monitoring endothelium-mediated changes in the digital pulse waveform, known as the Peripheral Arterial Tone (PAT) signal.
Metabolic effects (n=12) | up to 24 hours
  Additionally, 12 participants will be asked to collect a 24-hour urine specimen at two intervals (0-8 h and 8-24 h) the first day of each intervention, following the treatment ingestion (n=12).

SECONDARY OUTCOMES:
changes in glucose profile | change from baseline at 4 weeks
  Glucose will be determined by enzymatic methods (PENTRA 400).
changes in lipid profile | change from baseline at 4 weeks
  total-cholesterol will be determined by enzymatic methods (PENTRA 400).
changes in lipid profile | change from baseline at 4 weeks
  HDL-cholesterol will be determined by enzymatic methods (PENTRA 400).
changes in lipid profile | change from baseline at 4 weeks
  Triglycerides will be determined by enzymatic methods (PENTRA 400).
changes in lipid profile | change from baseline at 4 weeks
  LDL-cholesterol concentrations will be calculated with the Friedewald equation.
changes in oxidation profile | change from baseline at 4 weeks
  plasma oxidized LDL in urine will be measured by ELISA methods.
changes in inflammation enzymes | change from baseline at 4 weeks
  High sensitivity C-reactive protein (CRP) (immunoturbidimetry) in plasma by high sensitivity enzyme-immunoassays (ELISAs)
change in endothelial function | change from baseline endothelial function at 4 weeks
  Nitric oxide (NO) plasma concentrations will be measured through nitrates/nitrites ratio by colorimetry and those of Endothelin-1 by ELISA (both techniques from Cayman Chem. Co., Ann Arbor, USA).
Alcohol biomarker | change from baseline at 4 weeks
  Ethyl glucuronide in urine by Thermo Scientific Ethyl Glucuronide Enzyme Immunoassay.
Gene expression | change from baseline at 4 weeks
  Microfluidic cards (TaqMan® Gene Expression Array Microfluidic Card, 32.1 format, Applied Biosystems), 30 genes related with endothelial function and inflammation of a sub-sample of 30 subjects (15 by gender) will be determined in peripheral blood mononucleated cell (PBMC).

OTHER OUTCOMES:
Liver function test | through study completion, an average of 6 months
  Determination of liver transaminases (AST and ALT) as biomarkers of liver function in order to control liver damage as a result of alcohol administration

CONTACTS AND LOCATIONS:
Overall Officials: Rafael De la Torre Fornell, Pharm, PhD, Principal Investigator — IMIM-Hospital del Mar Medical Research Institute
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain